CLINICAL TRIAL: NCT00612820
Title: An 8 Day, Randomised, Double Blind, 3-way Crossover Trial of Repeat Doses of Intranasal GSK256066 and Fluticasone Propionate in the Vienna Challenge Chamber in Subjects With Seasonal Allergic Rhinitis (SAR)
Brief Title: A Phase II Study Evaluating Intranasal GSK256066 and Fluticasone Propionate in Subjects With Seasonal Allergic Rhinitis (SAR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IPR110723
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Vienna Challenge Chamber; Seasonal Allergic Rhinitis,
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — 6-((3-((dimethylamino)carbonyl)phenyl)sulfonyl)-8-methyl-4-((3-methyloxyphenyl)amino)-3-quinolinecarboxamide; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK256066 — 200mcg bd,
Drug: fluticasone propionate — 200mcg od,100mcg bd
  Other Names: GSK256066

SUMMARY:
This is an 8 day, randomised, double blind, 3-way crossover trial of repeat doses of intranasal GSK256066 and fluticasone propionate in the Vienna Challenge Chamber in subjects with seasonal allergic rhinitis (SAR). Approximately 60 subjects will be selected for enrolment with the intention of acquiring at least 48 evaluable subjects. Laboratory safety assessments, 12-lead electrocardiograph (ECG), vital signs and adverse event enquiries will be made throughout the study. Nasal examination, symptom scores, nasal lavage, nasal scrape and allergen challenge assessments will also be performed at various time points throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* The subject is healthy. Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history (including family), physical examination, laboratory studies, and other tests.
* They aged 18 to 50 years inclusive.
* Body mass index less than 29.0 kg/m² with weight range of 55.0kg (females 50kg) to 95.0kg inclusive.
* They have a history of seasonal allergic rhinitis.
* They exhibit a moderate response to 1500 grass pollen grains/m3 after 2h in the Vienna Challenge Chamber, which is defined as a nasal symptom score of at least 6. (Nasal symptom score is the sum of obstruction, rhinorrhoea, itch and sneeze, each of which have been scored on a scale from 0 to 3).
* They have a positive skin prick test (wheal ³ 4mm) for grass pollen at or within the 12 months preceding the screening visit.
* They have a positive RAST (³ class 2) for grass pollen at or within the 12 months preceding the screening visit.
* They are current non-smokers who have not used any tobacco products in the 6 months preceding the screening visit with a pack history of £ 10 pack years.

Pack years = No of cigarettes smoked/day

* They must have a baseline FEV1>80% predicted and a baseline FEV1 (maximum recorded value)/FVC (maximum recorded value)>70% predicted (using the Standardized Lung Function Testing guidelines produced by European Community for Coal and Steel).
* There are no conditions or factors which would make the subject unlikely to be able to stay in the chamber for 4 hours.
* They are capable of giving informed consent which includes compliance with the requirements and restrictions listed in the consent form.
* They are available to complete all study measurements.

Exclusion Criteria:

* Pregnant or nursing females.
* Women of childbearing potential who are unwilling or unable to use an appropriate method of contraception, as outlined below, from at least two weeks prior to the first dose of study medication; and to continue until the final pregnancy test has been performed.
* On examination the subject is found to have any structural nasal abnormalities or nasal polyposis, a history of frequent nosebleeds, recent nasal surgery or recent (within 2weeks) or ongoing upper respiratory tract infection which in the Responsible Physician's opinion renders the subject unsuitable for participation in the study.
* Any respiratory disease other than mild stable asthma that is controlled with occasional use of as-needed short-acting beta-agonists and associated with normal lung function.
* The subject is likely to be unable to abstain from salbutamol use for 8 hours before a challenge.
* The subject has a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* The subject is concurrently participating in another clinical study or has participated in a study with an investigational product (new chemical entity) during the previous 4 months or in any clinical study during the previous month.
* The subject has a screening QTc(B) value >450msec, PQ interval outside the range 120 to 240msec or an ECG that is not suitable for QT measurements (e.g. poorly defined termination of the T-wave). In addition subjects will be excluded if they have a history of atrial and ventricular arrhythmia.
* A supine blood pressure that is persistently higher than 140/90 millimetres of mercury (mmHg) at screening.
* A supine mean heart rate outside the range 40-90 beats per minute (bpm) at screening.
* The subject has donated a unit of blood (450mL) within the previous 3 months or intends to donate within 3 months of completing the study.
* The subject is currently taking regular (or a course of) medication whether prescribed or not, including steroids, vitamins, and herbal remedies (e.g. St. John's Wort). Subjects are not permitted to take potent inhibitors of cytochrome P450 3A4 including macrolide antibiotics or azole anti-fungals due to potential for increased systemic exposure to fluticasone propionate. Paracetamol (£2g/day) and occasional as needed use of short-acting beta agonists is permitted.
* The subject has used prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (which ever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Sponsor the medication will not interfere with the study procedures or compromise subject safety.
* The subject had used oral, injectable or dermal steroids within 5 weeks or intranasal and/or inhaled steroids within 1 week of the screening visit.
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease*, haematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, bronchiectasis or pulmonary fibrosis).

  *subjects will require normal serum creatinine clearance values at screening [calculated from serum creatinine by a predicting equation using Cockcroft-Gualt formula]. If the creatinine clearance value is greater than the upper limit of normal as determined by the local laboratory reference range, the Investigator will determine whether this is a clinically significant finding that would preclude participation.
* The subject regularly drinks more than 28 units of alcohol in a week if male, or 21 units per week if female. One unit of alcohol is defined as a medium (125 ml) glass of wine, half a pint (250 ml) of beer or one measure (24 ml) of spirits.

The subject is at risk of non-compliance with the study procedures/restrictions.

The subject is infected with the Hepatitis B, Hepatitis C, or HIV.

* The subject has an elevated Troponin T above the normal range.
* The subject has an elevated CK-MB above the normal range. Contraception for females

Appropriate contraceptive methods for female subjects include:

• Abstinence. The lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication and to continue until the follow up visit.

One of the following methods is acceptable as the sole method of contraception if there is indisputable data that it is >99% effective otherwise it should be used with a barrier method (condom or occlusive cap (diaphragm or cervical/vault caps) used with spermicidal foam/gel/film/cream/suppository):

* Documented tubal ligation
* Documented placement of an intrauterine device (IUD) or intrauterine system (IUS)
* Condom and occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Investigate effect of repeat intranasal doses of fluticasone propionate alone vs. GSK256066 + fluticasone propionate on nasal symptoms of allergic rhinitis provoked by spending 4 hours in the Vienna Challenge Chamber after morning dosing on Day 2. | spending 4 hours in the Vienna Challenge Chamber after morning dosing on Day 2.

SECONDARY OUTCOMES:
•Nasal symptoms | provoked after Day 2 dose.
•Nasal symptoms | after Day 8 dose.
Eye and global symptoms, nasal obstruction and secretions | after Day 2 and 8 dose.
Weighted mean TNSS (sneeze, itch, rhinorrhoea and obstruction) | 1 to 4hours post morning dose period spent in the Vienna Challenge Chamber on Day 8.
Weighted mean eye symptom score (watery eyes, itchy eyes, red eyes) | over 1 to 4 hours on Day 2 and 8.
Weighted mean global symptom score (sneeze, itch, rhinorrhoea, obstruction, cough, itchy throat, itchy ears, watery eyes, itchy eyes and red eyes) | over 1 to 4 hours on Day 2 and 8.
Weighted mean nasal airflow resistance (measured using active anterior rhinomanometry) and secretion weight (measured by weighing tissues) | over 1 to 4 hours on Day 2 and 8.
Weighted mean components of TNSS (sneeze, itch, rhinorrhoea and obstruction) | over 1 to 4 hours on Day 2 and 8.
FEV1, ECGs, Vitals, AEs, and laboratory safety parameters.
Effect of GSK256066 on ribonucleic acid (RNA) levels indicative of PDE4 inhibition in nasal scrape samples and on protein biomarkers of PDE4 inhibition in lavage samples
Effect of fluticasone propionate on RNA levels indicative of glucocorticoid-provoked gene expression in nasal scrape samples and on glucocorticoid receptor (GR) translocation in lavage samples

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: IPR110723 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: IPR110723 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: IPR110723 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: IPR110723 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: IPR110723 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: IPR110723 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: IPR110723 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register